CLINICAL TRIAL: NCT01628614
Title: A Study of Intraocular Pressure (IOP) Reduction in Newly Diagnosed Patients With Primary Open Angle Glaucoma (POAG) or Ocular Hypertension (OHT)
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: MAF/AGN/OPH/GLA/028; AGN-EPI-2010-01 (Other: Allergan)
Record Dates: First submitted 2012-06-25; First posted 2012-06-27 (Estimated); Results first posted 2012-09-05 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-08

CONDITIONS: Glaucoma, Open-Angle; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- POAG or OHT: Patients with POAG or OHT. All care (including treatment and diagnostic procedures) provided is at the discretion of the participating physicians according to their clinical judgment and the local standard of medical care.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Standard of Care — Patients with POAG or OHT. All care (including treatment and diagnostic procedures) provided is at the discretion of the participating physicians according to their clinical judgment and the local standard of medical care.

SUMMARY:
This is an observational study and will evaluate IOP reduction in newly diagnosed patients with POAG or OHT. All care (including treatment and diagnostic procedures) provided is at the discretion of the participating physicians according to their clinical judgment and the local standard of medical care.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed with primary open angle glaucoma or ocular hypertension

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with primary open angle glaucoma or ocular hypertension
Sampling Method: Non-Probability Sample
Enrollment: 4812 (Actual)
Dates: Start 2010-11; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Barcelona, Spain

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | POAG or OHT
Started | 4812
Completed | 3037
Not Completed | 1775

BASELINE CHARACTERISTICS:
Arm/Group | POAG or OHT
Number analyzed (Participants) | 4812
Age Continuous [Mean (Standard Deviation); unit: Years]
  Evaluable (N=2647 patients) | 64.72 (12.03)
  Missing (N=2165 patients) | NA (NA) — Age missing; not obtained
Sex/Gender, Customized [Number; unit: Participants]
  Female | 1642
  Male | 1389
  Missing | 1781

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With a Reduction in Intraocular Pressure (IOP) ≥ 5mmHg From Baseline
Description: Percentage of patients with a reduction in IOP≥5 mmHg from baseline. IOP is a measurement of the fluid pressure inside the eye. The minimum reduction of 5 mmHg was evaluated in the eye with the highest pressure at the baseline visit.
Time Frame: Baseline, 14 Weeks
Population: Evaluable Patients: all patients who met the study entry criteria
Measure: Number; unit: Millimeters of Mercury (mmHg)
Arm/Group | POAG or OHT
Number analyzed (Participants) | 3037
Millimeters of Mercury (mmHg) | 75.9

2. Secondary Outcome: Percentage of Patients With an IOP Reduction ≥10% From Baseline
Description: Percentage of patients with an IOP reduction ≥10% from baseline. IOP is a measurement of the fluid pressure inside the eye. The minimum reduction of 10% was evaluated in the eye with the highest pressure at the baseline visit.
Time Frame: Baseline, 14 Weeks
Population: Evaluable Patients: all patients who met the study entry criteria
Measure: Number; unit: Percentage of Patients
Arm/Group | POAG or OHT
Number analyzed (Participants) | 3037
Percentage of Patients | 91.0

3. Secondary Outcome: Percentage of Patients With an IOP Reduction ≥20% From Baseline
Description: Percentage of patients with an IOP reduction ≥20% from baseline. IOP is a measurement of the fluid pressure inside the eye. The minimum reduction of 20% was evaluated in the eye with the highest pressure at the baseline visit.
Time Frame: Baseline, 14 Weeks
Population: Evaluable Patients: all patients who met the study entry criteria
Measure: Number; unit: Percentage of Patients
Arm/Group | POAG or OHT
Number analyzed (Participants) | 3037
Percentage of Patients | 70.8

ADVERSE EVENTS:
Description: SAEs and AEs were analyzed for evaluable patients.
Arm/Group | POAG or OHT
Serious Adverse Events (participants affected / at risk) | 0/3037
Other Adverse Events (participants affected / at risk) | 180/3037
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | POAG or OHT (N=3037)
Ocular Hyperaemia (Eye disorders) | 180

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No